CLINICAL TRIAL: NCT01326351
Title: Plantar Fasciitis: Pain Relief and Improvement of Foot Function With Prolotherapy
Brief Title: Prolotherapy for the Treatment of Plantar Fasciitis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Réseau de Santé Vitalité Health Network (Other)
Responsible Party: Dr. Richard Dumais/ Professor, Pain Clinic Director, Anesthetist and Chronic Pain Specialist, Réseau de santé Vitalité Health Network
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: prolo-2011
Record Dates: First submitted 2011-03-29; First posted 2011-03-30 (Estimated); Last update posted 2011-04-19 (Estimated); Status verified 2011-04

CONDITIONS: Plantar Fasciitis
MeSH Terms: conditions — Fasciitis, Plantar | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Regenerative Injection Therapy (Experimental)
  Interventions: Procedure: Regenerative injection therapy
- Dry needle (Sham Comparator)
  Interventions: Procedure: Dry needle injection
- Exercise (Active Comparator)
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Procedure: Regenerative injection therapy — Injection of 10cc of a 15% dextrose and 0.6% lidocaine solution free of epinephrine in one injection site (lateral infiltration of the plantar fascia). This injection will be performed following posterior tibial nerve blockade (injection of 10cc of 1% lidocaine and 0.25% bupivacaine solution free of epinephrine behind the posterior tibial artery). The intervention will be administered every three weeks until symptoms are alleviated for a maximum of 5 injection sessions. Furthermore, patients must perform an at-home exercise program 3 times a week for a total of 12 weeks. The exercise program consists of 3 stretching exercises, 1 muscle release exercise and 1 strengthening exercise.
  Arms: Regenerative Injection Therapy
Procedure: Dry needle injection — Injection of dry needle in one injection site (lateral infiltration of the plantar fascia). This injection will be performed following posterior tibial nerve blockade(injection of 10cc of 1% lidocaine and 0.25% bupivacaine solution free of epinephrine behind the posterior tibial artery). The intervention will be administered every three weeks until symptoms are alleviated for a maximum of 5 injection sessions. Furthermore, patients must perform an at-home exercise program 3 times a week for a total of 12 weeks. The exercise program consists of 3 stretching exercises, 1 muscle release exercise and 1 strengthening exercise.
  Arms: Dry needle
Behavioral: Exercise — At-home exercise program that patients must perform 3 times a week for a total of 12 weeks. The exercise program consists of 3 stretching exercises, 1 muscle release exercise and 1 strengthening exercise.
  Arms: Exercise

SUMMARY:
The purpose of this study is to demonstrate that prolotherapy in conjunction with a physiotherapy program looking at reinforcing calf muscle and muscle of the plantar fascia, relieves pain and improves function of people suffering of plantar fasciitis, an inflammation of the plantar fascia, after basic treatment failure.

ELIGIBILITY:
Inclusion Criteria:

* have a diagnosis of Plantar Fasciitis
* experience pain in the plantar fascia for more than 6 months
* be capable to understand and execute physiotherapy exercises

Exclusion Criteria:

* previous operation of the plantar fascia
* deformation of the foot (congenital or acquired)
* presence or suspicion of infection of the skin at the site where the injection will occur
* history of systemic diseases capable of inducing pain or sensitivity to the feet (seronegative arthritis, diabetes, fibromyalgia, etc.)
* abnormal coagulation
* allergy to lidocaine and/or marcaine
* pregnancy
* lumbar, hip or knee pain

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-05; Primary Completion 2012-02 (Estimated); Study Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
Assessment of pain and function of the affected foot during the course of treatment | Every 3 weeks from week 0 to 36
  The Maryland Foot Score questionnaire will be used. This questionnaire assesses pain and function of injured foot using a summated rating scale of 10 questions.

SECONDARY OUTCOMES:
Assessment of pain intensity and pain-related function impairment during the course of treatment | Every 3 weeks from week 0 to 36
  The Brief Pain Inventory (short form) will be administered to assess pain intensity and pain-related functional impairment (physical and emotional). Four items assess the intensity of current pain and pain at ils least, worst, and average during the past day on scales form 0 ("no pain") to 10 ("pain as bad as you can imagine"). Seven more items measure pain-related functional interference in different domains (general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life) rated from 0 ("does not interfere") to 10 ("interferes completely").

CONTACTS AND LOCATIONS:
Locations (1):
- Dr.-Georges-L.-Dumont University Hospital Centre, Moncton, New Brunswick, Canada